CLINICAL TRIAL: NCT02371681
Title: NexGen EBA Radiologic and Immunologic Biomarkers of Sterilizing Drug Activity in Tuberculosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 999915070; 15-I-N070
Record Dates: First submitted 2015-02-25; First posted 2015-02-26 (Estimated); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Pulmonary Tuberculosis
Keywords: Treatment-Response; Radiological Imaging; Biomarkers; Antitubercular Agents; Log-CFU Reduction
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — Therapeutics; Specimen Handling

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): TB drugs
  Interventions: Drug: Treatment; Radiation: PET/CT Scan; Procedure: Sample Collection

INTERVENTIONS:
Drug: Treatment — Different Drug combinations
Radiation: PET/CT Scan — PET/CT Scans
Procedure: Sample Collection — Sample Collection

SUMMARY:
Background:

- Tuberculosis (TB) is a lung infection caused by bacteria. When people with TB cough, they may spread these bacteria. Researchers are looking for new TB medicines. They want to find a faster way to tell if a drug might combat TB.

Objective:

- To learn the effect of different anti-TB drugs on microbiological, radiographic and immunologic markers in people with TB.

Eligibility:

- Adults age 18-65 who weigh 30-90 kg and have common TB bacteria that can be treated with common TB medicines.

Design:

* Participants will be admitted to the hospital for screening. They will have medical history, physical exam, and chest radiograph. They will give blood, urine, and sputum samples.
* Participants will be put in 1 of 8 groups.
* Participants will get one or a combination of TB medicines daily for about 14 days.
* Each day, participants:
* Will discuss side effects.
* May have a physical exam.
* Will spit mucus into a cup. They may breathe in saline water through a nebulizer to make them cough.
* Participants will have blood taken 3-4 times during the study
* Participants will have 2-3 Fluorodeoxyglucose Positron Emission Tomography/Computed Tomography (FDG-PET/CT) scans. FDG is a radioactive sugar molecule which helps measure TB disease in the lungs. It will be injected into a vein. Participants will lie in a scanner that takes pictures.
* Around study day 14, participants will leave the hospital. They will be referred to a local TB clinic. There they will get the standard 4 TB medicines. Those in group 8 will already be on these medicines and will have another FDG-PET/CT on day 28.
* Participants will be in the study for up to 28 days.

DETAILED DESCRIPTION:
Early bactericidal activity (EBA), which measures decline in serial sputum colony forming unit (CFU) counts over the first 2-14 days of treatment, has been used extensively as a means of initially evaluating the potency of individual or combinations of antituberculous agents. This approach is endorsed by the Global Alliance for TB Drug Development and the US FDA. However, EBA seems to correlate poorly with the relative ability of an agent to prevent relapse and produce a durable cure (often referred to as sterilizing activity ). The reasons for this discrepancy may have to do with a limitation of sputum measurements to capture populations that persist beyond airway surfaces in discrete lesions such as granulomas, nodules, or cavities. The elimination of these persistent populations depend on the pharmacodynamic properties of a regimen and may be better captured by biologic and functional markers that can reflect dynamic treatment effects within these relevant host environments.

Recent studies of the response to TB chemotherapy have identified promising new biomarkers of sterilization in 2 areas. First, immunologic changes appear to have potential in small subject cohorts to predict sterilizing cure within 1 month after commencing treatment. Second, 18F-FDG PET/CT has been used in tuberculosis as a qualitative means of assessing drug response in small case series at multiple time points, starting as early as 1 month. PET activity reflects uptake and phosphorylation of FDG by neutrophils and macrophages, and CT provides structural information on disease pathology. Hence, PET/CT data may offer additional insights into lesion-specific sterilizing activity. This study will add 18F-FDG PET/CT scans and immunological assays at 0, 2, and (in the HRZE arm) 4 weeks to standard EBA methodology using regimens containing isoniazid (INH [H]), rifampin (RIF [R]), pyrazinamide (PZA [Z]), moxifloxacin (MXF [M]), and ethambutol (EMB [E]). We hypothesize that drug regimens associated with higher sterilizing activity (e.g., containing rifampin or pyrazinamide) will show distinctive early cytokine and chemokine patterns and discrete, quantifiable changes on PET/CT in certain lesion types during the 2-week period, compared to drug regimens with poor sterilizing activity (e.g., containing isoniazid or moxifloxacin). Demonstration of such an association would provide rationale for including radiologic and immunologic analysis, alongside conventional EBA, in early phase clinical studies of novel drugs, and would also provide important new insights into the biology of human and bacterial responses to TB drugs.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age 18 to 65 years with body weight from 30 kg to 90 kg
  2. Sputum acid-fast bacilli (AFB) smear positive (at least 1+ on the WHO International Union Against Tuberculosis and Lung Disease scale)
  3. Likely able to produce approximately 10 mL of sputum per day
  4. Xpert MTB/RIF-confirmed M.tb
  5. Rifampin-sensitive pulmonary tuberculosis as indicated by Xpert MTB/RIF
  6. ALT <3X upper limit of normal, creatinine <2X upper limit of normal
  7. Willingness to have samples stored

EXCLUSION CRITERIA:

1. Clinically suspected disseminated TB or acuity of illness too much as deemed by clinicians
2. Has been treated for tuberculosis within the past 3 years
3. Treatment with agents known to have anti-tuberculosis activity (e.g., fluoroquinolones, linezolid) for any indications during the current episode of clinical illness or within 2 months prior to screening, whichever is longer
4. Cirrhosis or chronic kidney disease
5. Disease complications or concomitant illness that might compromise safety or the interpretation of trial endpoints, such as known diagnosis of chronic inflammatory condition (e.g., sarcoidosis, rheumatoid arthritis, and connective tissue disorder)
6. Use of immunosuppressive medications, such as TNF-alpha inhibitors or systemic or inhaled corticosteroids, within 2 weeks prior to screening
7. Subjects with diabetes, point of care HbA1c above 6.5, or random glucose over 200 mg/dL
8. Conditions which compromise the subject s ability to take or absorb oral drugs
9. Normal PA-Chest radiograph, determined during screening
10. Total lung (left or right) collapse on PA-Chest radiograph
11. HIV positive
12. Pregnant or breastfeeding
13. Any other condition that, in the responsible clinician s judgment, renders a subject too sick to safely tolerate 2 weeks study therapy
14. Any condition that constitutes a contraindication to any of the drugs to be used on any study arms

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2015-02-25 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-11-14 (Actual)

PRIMARY OUTCOMES:
To characterize, in the context of a standard EBA study, the effect of various antituberculosis drugs on radiographic and immunologic markers as measured by PET/CT and immunologic assays, in subjects with drug sensitive pulmonary tuberculosis wh... | 14 days
  A description of the individual markers that change over time is of interest to better understand both the markers and the effects of each treatment. A second analysis will focus on classification of whether a treatment arm includes: 1) only one agent ( singlet ), 2) only two agents (a doublet ), or 3) four agents (a quadruplet ).

SECONDARY OUTCOMES:
PET/CT Changes | 14 days
  Correlation of PET/CT changes with treatment response, microbiologic and immunologic outcomes
Rank order of drugs | 14 days
  Comparison of the rank order of drugs based upon bacteriologic, radiologic and immunologic features.

CONTACTS AND LOCATIONS:
Overall Officials: Clifton E Barry, Ph.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (2):
- South Africa (2):
  - Stellenbosch University, Faculty of Medicine and Health Sciences, Cape Town
  - TASK Applied Sciences, Cape Town

REFERENCES:
- [Background] Dartois V, Barry CE. Clinical pharmacology and lesion penetrating properties of second- and third-line antituberculous agents used in the management of multidrug-resistant (MDR) and extensively-drug resistant (XDR) tuberculosis. Curr Clin Pharmacol. 2010 May;5(2):96-114. doi: 10.2174/157488410791110797. PMID 20156156
- [Background] Goo JM, Im JG, Do KH, Yeo JS, Seo JB, Kim HY, Chung JK. Pulmonary tuberculoma evaluated by means of FDG PET: findings in 10 cases. Radiology. 2000 Jul;216(1):117-21. doi: 10.1148/radiology.216.1.r00jl19117. PMID 10887236
- [Background] Jindani A, Dore CJ, Mitchison DA. Bactericidal and sterilizing activities of antituberculosis drugs during the first 14 days. Am J Respir Crit Care Med. 2003 May 15;167(10):1348-54. doi: 10.1164/rccm.200210-1125OC. Epub 2003 Jan 6. PMID 12519740
- [Derived] Jones A, Saini J, Kriel B, Via LE, Cai Y, Allies D, Hanna D, Hermann D, Loxton AG, Walzl G, Diacon AH, Romero K, Higashiyama R, Liu Y, Berg A. Sputum lipoarabinomannan (LAM) as a biomarker to determine sputum mycobacterial load: exploratory and model-based analyses of integrated data from four cohorts. BMC Infect Dis. 2022 Apr 2;22(1):327. doi: 10.1186/s12879-022-07308-3. PMID 35366820